CLINICAL TRIAL: NCT02195102
Title: Evaluation of Clinical Outcomes of Transcatheter Aortic Valve Replacement in the Asian Population The Asian Pacific TAVI Multicenter Registry A MULTICENTER, OBSERVATIONAL STUDY
Brief Title: The Asian Pacific TAVR Multicenter Registry
Acronym: AP TAVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Michael Kang-Yin Lee, MD (Other)
Collaborators: Asan Medical Center (Other); Cardiovascular Clinical Research (Industry)
Responsible Party: Sponsor-Investigator, Michael Kang-Yin Lee, MD, MD, Queen Elizabeth Hospital, Hong Kong
Organization: Queen Elizabeth Hospital, Hong Kong (Other)
Other Study IDs: AMCCV 2013-12
Record Dates: First submitted 2014-07-11; First posted 2014-07-21 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Aortic Valve Stenosis
Keywords: transcatheter aortic valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- transcatheter aortic valve Replacement: Patients with symptomatic severe aortic stenosis who are not candidates for surgical aortic valve replacement because of coexisting illnesses.
  Interventions: Device: Transcatheter aortic valve Replacement

INTERVENTIONS:
Device: Transcatheter aortic valve Replacement

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of transcatheter aortic valve Replacement (TAVR) in the Asian Pacific population

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic severe aortic stenosis who are not candidates for surgical aortic valve replacement because of coexisting illnesses.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who had undergone transcatheter aortic valve replacement on the basis of inclusion criteria were prospectively&retrospectively included in the registry
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-12; Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 1 month
Death from any cause | 6 months
Death from any cause | 1 year
Death from any cause | 2 years
Death from any cause | 3 years
Death from any cause | 4 years
Death from any cause | 5 years

SECONDARY OUTCOMES:
Death from cardiac cause | 1 month
Death from cardiac cause | 6 months
Death from cardiac cause | 1 year
Death from cardiac cause | 2 years
Death from cardiac cause | 3 years
Death from cardiac cause | 4 years
Death from cardiac cause | 5 years
Stroke | 1 month
Stroke | 6 months
Stroke | 1 year
Stroke | 2 years
Stroke | 3 years
Stroke | 4 years
Stroke | 5 years
Myocardial infarction | 1 month
Myocardial infarction | 6 months
Myocardial infarction | 1 year
Myocardial infarction | 2 years
Myocardial infarction | 3 years
Myocardial infarction | 4 years
Myocardial infarction | 5 years
Repeat hospitalization | 1 month
Repeat hospitalization | 6 months
Repeat hospitalization | 1 year
Repeat hospitalization | 2 years
Repeat hospitalization | 3 years
Repeat hospitalization | 4 years
Repeat hospitalization | 5 years
Acute kidney injury | 1 month
Acute kidney injury | 6 months
Acute kidney injury | 1 year
Acute kidney injury | 2 years
Acute kidney injury | 3 years
Acute kidney injury | 4 years
Acute kidney injury | 5 years
Vascular complication | 1 month
Vascular complication | 6 months
Vascular complication | 1 year
Vascular complication | 2 years
Vascular complication | 3 years
Vascular complication | 4 years
Vascular complication | 5 years
Bleeding events | 1 month
Bleeding events | 6 months
Bleeding events | 1 year
Bleeding events | 2 years
Bleeding events | 3 years
Bleeding events | 4 years
Bleeding events | 5 years
Device success | 1 month
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 6 months
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 1 year
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 2 years
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 3 years
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 4 years
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Device success | 5 years
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, PhD, Principal Investigator — Asan Medical Center, Republic of Korea; Edgar L.W. Tay, MD, Principal Investigator — National University Heart Center (National University Health System), Singapore; Machael Kang-Yin Lee, MD, Principal Investigator — Queen Elizabeth Hospital, HongKong
Locations (10):
- China (2):
  - Queen Elizabeth Hospital, Hong Kong
  - Nanjing 1st Hospital, Nanjing
- Shonan Kamakura General Hospital, Kamakura, Japan
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- St. Luke's Medical Center, Bonifacio, Philippines
- Singapore (2):
  - National Heart Centre of Singapore, Singapore
  - National University Heart Centre, Singapore
- Asan Medical Center, Seoul, South Korea
- National Taiwan University, Taipei, Taiwan
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand